CLINICAL TRIAL: NCT05638893
Title: Metformin as Adjuvant Therapy in Obese Knee Osteoarthritis Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amany Abd Elaal Mohamed Aiad, pharmacist, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Metformin knee osteoarthritis
Record Dates: First submitted 2022-11-28; First posted 2022-12-06 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Knee Osteoarthritis
Keywords: Metformin; knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Metformin; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Experimental): Placebo tablet twice daily + celecoxib 200mg capsule once daily for 12 weeks.
  Interventions: Drug: Placebo Tablet
- Metformin group (Experimental): Metformin 500mg tablet twice daily + celecoxib 200mg capsule once daily for 12 weeks.
  Interventions: Drug: Metformin Hcl 500Mg Tab

INTERVENTIONS:
Drug: Placebo Tablet — Placebo (tablet/12hr) + celecoxib (200mg/day) for three months.
  Arms: Placebo group
Drug: Metformin Hcl 500Mg Tab — Metformin (500mg/12hr) + celecoxib (200mg/day) for three months.
  Other Names: Cidophage 500mg Oral Tablet
  Arms: Metformin group

SUMMARY:
This study aims to evaluate the possible efficacy and safety of addition of metformin to celecoxib in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Metformin is a safe, well-tolerated oral biguanide widely used as first-line therapy for type 2 diabetes for over 50 years. In addition to its glucose-lowering effects, metformin modulates inflammatory and metabolic factors resulting in weight loss and reduced inflammation and plasma lipids. Data from animal studies suggest that metformin could limit OA development and progression, possibly through activating AMPK.

Retrospective cohort study of participants with OA and type 2 diabetes reported that patients receiving a combination of cyclooxygenase-2 inhibitors and metformin therapy had a lower risk of joint replacement than those receiving cyclooxygenase-2 inhibitors alone .

These findings shed light on possible therapeutic potential of metformin in treatment of OA.

ELIGIBILITY:
Inclusion Criteria:

* Patients have symptomatic and radiological evidence of OA in one or both knee joints.
* Age ≥ 45 years.
* Both obese male and female will be included (BMI ≥ 30 kg/m²).

Exclusion Criteria:

* Patients with inflammatory rheumatic diseases, crystal deposition arthritis or infection-induced OA.
* Patient with hypertension or diabetes mellitus.
* Patient with hepatic or renal impairment.
* Patients who have active peptic ulcer.
* Patients with positive malignancy.
* Steroid injection into the affected knee joint within 3 months of recruitment for the study.
* Pregnant or lactating female patients.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-03-12 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 12 weeks
  Measure change in Western Ontario and McMaster Universities Arthritis Index (WOMAC) at baseline and after 12weeks of treatment.
Weight (Kg) | 12 weeks
  Measure change in weight in kilograms at baseline and after 12weeks of treatment.

SECONDARY OUTCOMES:
Cartilage Oligomeric Matrix Protein (COMP) | 12 weeks
  Measure change in Cartilage Oligomeric Matrix Protein (COMP) serum level at baseline and after 12weeks of treatment.
C-terminal crosslinked telopeptide of type I collagen (CTX-1) | 12 weeks
  Measure change in C-terminal crosslinked telopeptide of type I collagen (CTX-1) serum level at baseline and after 12weeks of treatment.
Interleukin 1-beta (IL-1β) | 12 weeks
  Measure change in Interleukin 1-beta (IL-1β) serum level at baseline and after 12weeks of treatment.
Adverse drug events | 12 weeks
  side effects

CONTACTS AND LOCATIONS:
Overall Officials: Sahar M El-Haggar, Professor, Study Chair — Tanta University; Amal M El-Barbary, Professor, Study Chair — Tanta University
Locations (1):
- Tanta university, Tanta, Gharbia Governorate, Egypt

REFERENCES:
- [Derived] Aiad AAE, El-Haggar SM, El-Barbary AM, El-Afify DR. Metformin as adjuvant therapy in obese knee osteoarthritis patients. Inflammopharmacology. 2024 Aug;32(4):2349-2359. doi: 10.1007/s10787-024-01495-y. Epub 2024 Jun 13. PMID 38869746